CLINICAL TRIAL: NCT06459895
Title: Biochemical Role of Long Non-coding RNA MALAT 1 and Serum Tumor Necrosis Factor Alpha in Bronchial Asthma Patients.
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Zainab Mahmoud Kadry, MD in Medical Biochemistry, Sohag University
Other Study IDs: Soh-Med-24-05-03PD
Record Dates: First submitted 2024-06-10; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples With DNA — Ten ml of blood was collected from patients by venipuncture. Samples were divided into two parts. The first part was added to EDTA (Ethylenediamine-tetra acetic acid) tube, until the extraction of RNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- diseased group: bronchial asthma diseased group
  Interventions: Diagnostic Test: Long non-coding MALAT1 gene expression assay:
- control group: healthy person
  Interventions: Diagnostic Test: Long non-coding MALAT1 gene expression assay:

INTERVENTIONS:
Diagnostic Test: Long non-coding MALAT1 gene expression assay: — RNA extraction (isolation from whole blood) II-Synthesis of CDNA from RNA by reverse transcription III-Gene expression assay by RT-PCR reaction

SUMMARY:
Bronchial asthma affects more than a quarter of a billion people worldwide. It is responsible for over 1000 deaths a day, of which the majority are preventable (Levy, 2015).

Asthma is a common heterogeneous disease characterized by chronic airway inflammation. It is defined by the history of variable respiratory symptoms, such as shortness of breath, chest tightness, wheezes, and cough, together with variable expiratory airflow limitation. Airflow limitation may later become persistent (GINA, 2023).

The diagnosis of asthma is based on the history of these characteristic symptoms and evidence of variable expiratory airflow limitation from bronchodilator reversibility testing or other tests (GINA, 2023).

ELIGIBILITY:
Inclusion Criteria:

* All patients were admitted to Sohag University Hospital, chest department DIAGNOSED AS BRONCHIAL ASTHMA

Exclusion Criteria:

* Patients with malignancies, major trauma or surgery, and acute or chronic infectious diseases were excluded.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study was case control had included 97 asthma patients and 97 healthy controls. The asthmatic patients will cautiously select from those attending the respiratory consultant clinics at Sohag University Hospital diagnosed with asthma (with no history of respiratory infections) PFT was performed with a spirometer (PHILIPS). The primary purpose of it was to confirm the diagnosis of asthma. Pre- and post-bronchodilator spirometer measurements will be performed in all study subjects and forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC) values and FEV1/FVC ratio will be
Sampling Method: Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Long non-coding MALAT1 gene expression assay: | 2 MONTHS
  Gene expression assay by RT-PCR reaction

SECONDARY OUTCOMES:
TNF-alpha | 2 MONTHS
  measured in serum by ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Background] Choi JP, Kim YS, Kim OY, Kim YM, Jeon SG, Roh TY, Park JS, Gho YS, Kim YK. TNF-alpha is a key mediator in the development of Th2 cell response to inhaled allergens induced by a viral PAMP double-stranded RNA. Allergy. 2012 Sep;67(9):1138-48. doi: 10.1111/j.1398-9995.2012.02871.x. Epub 2012 Jul 5. PMID 22765163
- [Background] Levy ML. The national review of asthma deaths: what did we learn and what needs to change? Breathe (Sheff). 2015 Mar;11(1):14-24. doi: 10.1183/20734735.008914. PMID 26306100
- [Background] Lee CG, Link H, Baluk P, Homer RJ, Chapoval S, Bhandari V, Kang MJ, Cohn L, Kim YK, McDonald DM, Elias JA. Vascular endothelial growth factor (VEGF) induces remodeling and enhances TH2-mediated sensitization and inflammation in the lung. Nat Med. 2004 Oct;10(10):1095-103. doi: 10.1038/nm1105. Epub 2004 Sep 19. PMID 15378055